CLINICAL TRIAL: NCT06149325
Title: Stimulate One Hand to Improve Tactile Perception on the Other
Acronym: HAND-HAND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 69HCL23_0913; 2023-A01994-41 (Other: ID-RCB)
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Post-stroke Sensory Deficits at the Hand
Keywords: Stroke; Sensory deficits; RSS
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The study is a comparative study, to show that the administration of RSS stimulation leads to a better performance compared to the administration of Sham stimulation (control). The participant's performance after receiving Sham stimulation will be unchanged compared to the baseline performance measured before the stimulation. On the contrary, participant's performance after receiving RSS stimulation will show a considerable improvement compared to the baseline performance, proving the superiority of RSS stimulation over the control. The study has a cross-over design, where each participant receives both stimulations, on different days. The two stimulations will be administered in a randomized order across participants, and in double-blind.
Who Masked: Participant, Investigator
Masking Description: Experimenter 2 will be in charge of the randomization. He will establish a randomization list through Excel and assign to each patient one of the two possible order (Day 1 RSS / Day 2 Sham OR Day 1 Sham / Day 2 RSS). This Excel will be protected through a password and kept in the CRNL server. He will then fill the envelopes with the order assigned by the randomization list and seal them. Each envelope is assigned an inclusion number.
  On the inclusion visit (J0), once the consent form is signed, the sealed envelope will be kept in the medical file of the patient. On the first visit (J1). Experimenter 1 will assess the performance of the patient through the tactile and motor tests, while the Exp2 will be in charge of applying the stimulation.
  Once Exp1 finished doing the tactile and motor tasks, she will leave the room and Exp2 will enter in the room, open the sealed envelope and apply the stimulation. He will stay in the room with the patient during the stimulation duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repetitive somatosensory stimulation (RSS), then SHAM (Experimental): Adult patients suffering from post-stroke sensory deficits at the hand. Each participant will participate to the study on two different days, at least a week apart from each other. The length of the experimental session on these two days will be the same: 2 hours in the morning, to perform Pre-evaluation of the tactile acuity, absolute detection, overall hand functionality and manual dexterity, and 3 hours in the afternoon, including 45 minutes of stimulation (RSS or Sham) and 2 hours of Post-evaluation of the tactile acuity, absolute detection, overall hand functionality and manual dexterity. In total, the length of the participation of each patient will be of 10 hours, spread on two days.
  Interventions: Procedure: Repetitive somatosensory stimulation (RSS); Procedure: Sham Repetitive somatosensory stimulation (RSS)
- Sham Repetitive somatosensory stimulation (RSS), then RSS (Experimental): Adult patients suffering from post-stroke sensory deficits at the hand. Each participant will participate to the study on two different days, at least a week apart from each other. The length of the experimental session on these two days will be the same: 2 hours in the morning, to perform Pre-evaluation of the tactile acuity, absolute detection, overall hand functionality and manual dexterity, and 3 hours in the afternoon, including 45 minutes of stimulation (RSS or Sham) and 2 hours of Post-evaluation of the tactile acuity, absolute detection, overall hand functionality and manual dexterity. In total, the length of the participation of each patient will be of 10 hours, spread on two days.
  Interventions: Procedure: Repetitive somatosensory stimulation (RSS); Procedure: Sham Repetitive somatosensory stimulation (RSS)

INTERVENTIONS:
Procedure: Repetitive somatosensory stimulation (RSS) — Tactile stimuli on the index finger of the intact hand, for a duration of 45 minutes
Procedure: Sham Repetitive somatosensory stimulation (RSS) — Tactile stimuli on the index finger of the intact hand, for a duration of 4 minutes spread over 45 minutes in 6 blocks of 40 seconds

SUMMARY:
The study is a comparative study, to show that the administration of RSS stimulation on one hand compared to the administration of strategy Sham stimulation, results in an temporary improvement in the tactile acuity of the other hand in patients with tactile acuity impairment of the hand due to stroke.

ELIGIBILITY:
* Inclusion Criteria:

  * Age: 30-80 years old
  * Patients with diagnosis of unilateral (both right and left) ischemic or hemorrhagic stroke
  * Stroke event dates at least 3 months before the date of inclusion to the study
  * Severe-to-mild sensory loss at the fingers of the hand contralateral to the stroke lesion (affected hand)
  * Capacity to provide written consent
  * Affiliation to a social security scheme
* Non inclusion Criteria * :

  * Sensory impairment attributable to diabetes history, peripheral vascular disease or neuropathy
  * Severe speech disorder, global aphasia and/or cognitive impairment
  * Multiple stroke events
  * Bilateral stroke event
  * History of neurological or psychiatric illness
  * Other experimental procedure is forbidden during the weeks where the study is performed
  * Pregnant, parturient and lactating women
  * Persons deprived of their liberty
  * Adult persons subject to a legal protection measure: guardianship, curatorship
  * Persons in psychiatric care
  * Congenital or acquired malformation/injury of the test fingers
  * Impossibility to maintain hand position necessary for the tests due to severe spasticity

Exclusion Criteria:

• Severe impairment of the sensibility of the index finger of the spared hand preventing the administration of the RSS

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Tactile acuity : composite of 2point discrimination test (2PDT) and Absolute threshold detection test after 45minutes of RSS | Immediate after the 45 minutes of RSS
  To show that RSS applied for 45 minutes on the index finger of the spared hand in stroke patients suffering from sensory deficits improves their tactile sensitivity on the affected (unstimulated) hand, measured in terms of improved spatial discrimination and/or improved absolute detection.

SECONDARY OUTCOMES:
Jebsen-Taylor hand function test (JTHFT) | Immediate after the 45 minutes of RSS
  Overall functionality of the hand, especially with regard to handling objects
Manual dexterity Pegboard test | Immediate after the 45 minutes of RSS
  Assessment of manual dexterity of the affected unstimulated hand (as well as of the spared hand)

CONTACTS AND LOCATIONS:
Locations (1):
- Groupement Hospitalier du Sud - Hôpital Henry Gabrielle, Saint-Genis-Laval, France

IPD SHARING:
Plan to Share IPD: Undecided